CLINICAL TRIAL: NCT06129513
Title: The Effect of a Novel Plant-blend Protein Isolate on Post-exercise Myofibrillar Protein Synthesis When Compared to Whey Protein in Healthy Young Adults
Brief Title: The Effect of a Plant-blend Protein Isolate on Post-exercise Myofibrillar Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-02-02-B-02
Record Dates: First submitted 2023-09-20; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Muscle Metabolism
Keywords: Myofibrillar Protein Synthesis; Resistance Exercise; Plant Protein; Stable Isotopes
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey protein isolate (Active Comparator): Following a bout of bilateral resistance exercise, participants will ingest 32 g protein from whey protein isolate
  Interventions: Behavioral: Bilateral resistance exercise; Dietary Supplement: Whey protein
- Plant-blend isolate (Experimental): Following a bout of bilateral resistance exercise, participants will ingest 32 g protein from a novel plant-blend protein isolate
  Interventions: Behavioral: Bilateral resistance exercise; Dietary Supplement: Plant-blend protein

INTERVENTIONS:
Behavioral: Bilateral resistance exercise — A bout of bilateral resistance exercise consisting of barbell back squat, leg leg press and leg extension
Dietary Supplement: Whey protein — Following execution of bilateral resistance exercise, participants will ingest 32 g protein from whey protein isolate
  Arms: Whey protein isolate
Dietary Supplement: Plant-blend protein — Following execution of bilateral resistance exercise, participants will ingest 32 g protein from plant-blend protein isolate
  Arms: Plant-blend isolate

SUMMARY:
Dietary protein ingestion is required to maximise the anabolic response during the recovery from resistance exercise. Whey protein is considered the optimal dietary strategy to maximise post-exercise muscle protein synthesis, but animal-protein production and consumption is associated with growing environmental and ethical concerns. Plant-based protein sources are considered of lesser anabolic quality than isonitrogenous boluses of animal-derived protein attributed to, at least in part, deficiencies in key essential amino acid. Blending different protein sources may overcome amino acid deficiencies and potentiate the post-exercise anabolic response. In the present study the investigators assessed the post-exercise muscle protein synthetic response following the ingestion of a novel plant-based protein isolate when compared with an isonitrogenous bolus of whey protein in healthy young, resistance trained women and men.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 - 30
* Resistance trained (>3 times per week structured resistance exercise training for at least 3 months)

Exclusion Criteria:

* Any metabolic impairment
* Any cardiovascular impairment
* Smoking
* Lactose intolerance
* Allergies to products containing dairy, meat or nuts
* Prescribed intake of over the counter pharmaceuticals

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Post-exercise myofibrillar protein synthesis following protein ingestion | 4 hours
  The fractional synthetic rate of myofibrillar proteins

SECONDARY OUTCOMES:
Post-exercise myofibrillar protein synthesis during the early postprandial period | 2 hours
  The fractional synthetic rate of myofibrillar proteins
Post-exercise myofibrillar protein synthesis during the late postprandial period | 2 hours
  The fractional synthetic rate of myofibrillar proteins
Plasma amino acid response | 4 hours
  Post-exercise and postprandial change in plasma amino acid concentrations and availability
Serum insulin response | 4 hours
  Post-exercise and postprandial change in serum insulin concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, United Kingdom

REFERENCES:
- [Derived] VAN DER Heijden I, Monteyne AJ, West S, Morton JP, Langan-Evans C, Hearris MA, Abdelrahman DR, Murton AJ, Stephens FB, Wall BT. Plant Protein Blend Ingestion Stimulates Postexercise Myofibrillar Protein Synthesis Rates Equivalently to Whey in Resistance-Trained Adults. Med Sci Sports Exerc. 2024 Aug 1;56(8):1467-1479. doi: 10.1249/MSS.0000000000003432. Epub 2024 Mar 23. PMID 38537270